CLINICAL TRIAL: NCT03793101
Title: Analysis of Quality of Vision and Eye Tissue Complications in Patients Operated With Biaxial Microincision Surgery Technique.
Brief Title: Biaxial Microincision Cataract Surgery Technique
Acronym: BiMICS14vs18
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Eyemed Centrum Okulistyczne (Other)
Responsible Party: Principal Investigator, Paweł Klonowski, Dr Paweł Klonowski Medical Director, Eyemed Centrum Okulistyczne
Other Study IDs: EYE0001
Record Dates: First submitted 2018-12-29; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Cataract Senile
Keywords: BiMICS, biaxial cataract surgery, SIA,diabetes mellitus,

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BiMICS 1.4: Group 1.4 - Patients operated with 1.4 mm BiMICS technique
  Interventions: Procedure: BiMICS
- BiMICS 1.8: Group 1.8 - Patients operated with 1.8 mm BiMICS technique
  Interventions: Procedure: BiMICS

INTERVENTIONS:
Procedure: BiMICS — Biaxial microincision cataract surgery implies performing of 2 corneal incisions under 1.8mm, removal of the crystalline lens with the use of ultrasounds and implantation of the artificial intraocular lens.

SUMMARY:
To analyze and compare visual results, keratometry, SIA and HOAs outcomes of biaxial microincision cataract surgery in elderly population, including diabetic and non-diabetic patients.

DETAILED DESCRIPTION:
Modern trends in cataract surgery is the bimanual MICS technique. MICS significant development for 15 years gives possibility to implant the intraocular lens by 1.4mm incision. This is not only a change in surgery technique, but it is a significant progress in safety and quality post-operative results. Bimanual cataract MICS technique gives the opportunity to reduce width of the corneal incision more than 40% comparing to the standard coaxial cataract surgery by use dedicated MICS IOL's. This allows to perform less traumatic surgery and provides the opportunity for fast visual rehabilitation from the first week after cataract surgery. The possibility of using multifocal and toric intraocular lenses in MICS technique fully meet the requirements of modern refractive intraocular surgery.

ELIGIBILITY:
Inclusion Criteria:

1.Clinical diagnose of senile cataract.

Exclusion Criteria:

1. Eye trauma in anamnesis.
2. Eye surgery in anamnesis.
3. Corneal surgery in anamnesis.
4. Corneal irregular astigmatism.
5. Corneal ectasia.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 3 months
  Snellen charts, EDTRS charts

SECONDARY OUTCOMES:
Keratometry | 3 months
  Diopters
Surgically Induced Astigmatism, SIA | 3 months
  Diopters
Higher Order Aberrations, HOAs | 3 months
  Micrones
Corneal Incision thickness | 3 nmonths
  Micrones

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Klonowski, MD, Principal Investigator — Eyemed Centrum Okulistyczne
Locations (1):
- Eyemed Centrum Okulistyczne, Lublin, Poland

IPD SHARING:
Plan to Share IPD: Yes
UCVA, BCVA, SIA, HOAs, Corneal Incision thickness
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from August 2019 until December 2020
Access Criteria: only on request
URL: http://eyemed.pl

REFERENCES:
- See also: MICS and Incise IOL — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6153898/
- Available data/document: Clinical Study Report — http://eyemed.pl